CLINICAL TRIAL: NCT03486860
Title: A Multi-Method Early Intervention Program for Inhibited and Anxious Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Andrea Chronis-Tuscano, Professor, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH083832 (NIH)
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Behavioral Inhibition; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Turtle Program (Experimental): The Turtle Program involves a child social and emotional skills group (Social Skills Facilitated Play) and a modification of Parent-Child Interaction Therapy in which parents are provided in-vivo coaching in following their children's lead and encouraging approach behaviors within the peer context. The child group provides a forum of same-age peers to learn to develop social and emotion regulation skills. The Turtle Program is administered over an 8-week period.
  Interventions: Behavioral: Turtle Program
- Waitlist Control (Other): Untreated comparison group during the study, received parent psychoeducation intervention after the active treatment group.
  Interventions: Behavioral: Parent Psychoeducation

INTERVENTIONS:
Behavioral: Parent Psychoeducation — 6-session parent psychoeducation group on child anxiety, following their children's lead, and encouraging approach behaviors.
  Arms: Waitlist Control
Behavioral: Turtle Program — The Turtle Program involves a child social and emotional skills group (Social Skills Facilitated Play) and a modification of Parent-Child Interaction Therapy in which parents are provided in-vivo coaching in following their children's lead and encouraging approach behaviors within the peer context. The child group provides a forum of same-age peers to learn to develop social and emotion regulation skills. The Turtle Program is administered over an 8-week period.
  Arms: Turtle Program

SUMMARY:
This project aims to develop and evaluate a novel early intervention program that targets the specific risk factors implicated in the development and persistence of shyness, social reticence, and withdrawal in children. The project includes a program development phase, Phase I (pilot test of full study procedures using developed treatment protocol), and Phase II (randomized controlled trial/RCT). Outcomes that will be assessed include change in child behavioral inhibition and parenting, using parent and teacher reports and observational data. Families are assessed at three time points: baseline, post-treatment (or at approximately 8 weeks for the control group), and 2 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Child must be attending preschool; child must score within top 15% on parent-rated Behavioral Inhibition Questionnaire; child has a biological parent with at least 50% physical custody who consents to participate

Exclusion Criteria:

* Child has a diagnosis of pervasive developmental disorder or mental retardation; child scores above clinical cutoff on Social Communication Questionnaire; child is currently receiving treatment for anxiety

Ages: 42 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2012-11-30 (Actual); Study Completion 2012-11-30 (Actual)

PRIMARY OUTCOMES:
Change in child anxiety disorder symptoms | Pre-treatment (baseline), post-treatment (week 8), and 2-month follow-up
  Assessed with diagnostic interviews (Preschool Age Psychiatric Assessment) with parents

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Chronis-Tuscano, Ph.D., Principal Investigator — University of Maryland; Kenneth Rubin, Ph.D., Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, College Park, Maryland, United States